CLINICAL TRIAL: NCT07352384
Title: Evaluation of the Efficacy of Neuromodulation in the Control of Chronic Orofacial Pain: A Randomized Controlled Trial
Brief Title: Evaluation of the Efficacy of Neuromodulation in the Control of Chronic Orofacial Pain
Acronym: NeuroFace
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: University of Sao Paulo (Other); University of Aarhus (Other); Universidade Federal de Alfenas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEEM1660
Record Dates: First submitted 2025-11-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Orofacial Pain
Keywords: Transcranial Magnetic Stimulation (TMS); Transcranial Direct Current Stimulation (tDCS); Neuromodulation; Orofacial Pain; Chronic Pain
MeSH Terms: conditions — Facial Pain; Chronic Pain | interventions — Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This randomized, parallel-group, double-blind, sham-controlled interventional trial evaluates the efficacy of non-invasive neuromodulation (tDCS or TMS) in adults with chronic orofacial pain. Participants are allocated 1:1 to active or sham stimulation through a computer-generated randomization sequence. The study includes baseline assessments, a 2-week intervention period, and post-treatment evaluations using validated clinical and functional measures. Blinding is maintained for participants and outcome assessors, with stimulation operators following standardized procedures to prevent unblinding. This design allows a controlled comparison of pain reduction, functional improvement, and safety between groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and outcome assessors are blinded to group assignment. Active and sham neuromodulation follow identical procedures, session durations, and device setups to maintain blinding. Stimulation operators administer the assigned condition but do not participate in assessments or data analysis to prevent disclosure of allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Neuromodulation (Active Comparator): Participants assigned to this arm receive active neuromodulation using either transcranial direct current stimulation (tDCS) or transcranial magnetic stimulation (TMS), according to the study protocol. Stimulation parameters follow standardized therapeutic settings, including electrode/coil placement, intensity, and session duration. The intervention is delivered over a 2-week schedule. Active stimulation is designed to modulate cortical excitability and pain-related neural circuits.
  Interventions: Device: Active Neuromodulation (tDCS or TMS)
- Sham/Placebo Neuromodulation (Placebo Comparator): Participants in this arm receive sham (placebo) neuromodulation designed to mimic the sensory experience of tDCS or TMS without delivering effective stimulation. For tDCS, the device provides brief ramp-up/ramp-down current; for TMS, a sham coil or tilted coil reproduces sound and scalp sensation without inducing cortical effects. Procedures, duration, and interactions are identical to the active arm to maintain blinding.
  Interventions: Device: Sham Neuromodulation (tDCS or TMS)

INTERVENTIONS:
Device: Active Neuromodulation (tDCS or TMS) — Participants receive active non-invasive neuromodulation using either transcranial direct current stimulation (tDCS) or transcranial magnetic stimulation (TMS).
  For tDCS, stimulation is delivered with 35 cm² electrodes, 1-2 mA, for 20 minutes, with the anode placed over C3 or C4 contralateral to the pain side, for five consecutive sessions.
  For TMS, stimulation is delivered with a figure-of-eight coil targeting the motor cortex corresponding to the orofacial region, following established safety protocols (e.g., 10 sessions across two weeks).
  All procedures follow standardized therapeutic parameters aiming to modulate cortical excitability and reduce pain.
  Other Names: Active tDCS; Active TMS; Active neuromodulation therapy
  Arms: Active Neuromodulation
Device: Sham Neuromodulation (tDCS or TMS) — Participants receive sham stimulation designed to mimic the sensory experience of tDCS or TMS without producing physiological neuromodulatory effects.
  For tDCS, the device uses brief ramp-up/ramp-down currents to simulate tingling without active stimulation.
  For TMS, a sham coil or angled coil is used to reproduce acoustic and scalp sensations while preventing magnetic induction.
  Session duration, procedures, and interaction with the operator are identical to the active arm to maintain blinding integrity.
  Other Names: Sham tDCS; Sham TMS; Placebo neuromodulation
  Arms: Sham/Placebo Neuromodulation

SUMMARY:
Chronic orofacial pain significantly affects patients' quality of life, compromising essential functions such as chewing and speech. Although conventional treatments are available, many patients do not achieve adequate and lasting relief. This project investigates the effectiveness of neuromodulation techniques, namely transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS), as innovative therapeutic alternatives for the control of chronic orofacial pain.

The study will be conducted in adult patients diagnosed with orofacial pain. Participants will be divided into two groups: one group will receive active neuromodulation (tDCS or TMS) and the other a sham treatment (placebo). Sessions will take place daily over two weeks. Assessments will include pain intensity, pain pressure threshold, masticatory function, and bite strength, in order to observe any functional changes.

The group undergoing neuromodulation is expected to show a significant reduction in pain levels and improvements in quality of life compared to the placebo group. This study could support the adoption of neuromodulation as a complementary approach in the treatment of chronic orofacial pain, offering an effective and non-invasive alternative for patients who do not respond to conventional treatments.

DETAILED DESCRIPTION:
The study will be conducted at the University Clinic of the Egas Moniz School of Health and Science - Department of Orofacial Pain. The objective is to evaluate the effects of electrical and magnetic neuromodulation on different chronic pain conditions using standardized non-invasive brain stimulation protocols and validated clinical and functional assessment instruments.

Sample

Individuals with chronic low back pain (score between 40 and 80 on the Portuguese version of the Oswestry Disability Index) and chronic orofacial pain (score between 40 and 80 on the Portuguese version of the Manchester Orofacial Pain Disability Scale) will be selected.

For each chronic pain condition, 50 individuals will be enrolled and allocated into two groups: a control group and an intervention group.

Inclusion Criteria

Age between 18 and 75 years.

Diagnosis of chronic orofacial pain lasting longer than 3 months, confirmed by validated diagnostic criteria such as DC/TMD.

Initial Visual Analogue Scale (VAS) score ≥ 4.

Previous attempt of at least one conventional treatment with limited effectiveness.

Cognitive capacity sufficient to understand study procedures and provide informed consent.

Stable chronic pain medication regimen for at least four weeks prior to the intervention.

Exclusion Criteria

History of epilepsy, seizures, or other neurological conditions that contraindicate tDCS or TMS.

Presence of implanted medical devices, including pacemakers, cochlear implants, or other electronic/metallic devices in the head or neck region.

Pregnancy or breastfeeding.

Severe psychiatric disorders that may compromise adherence to study procedures.

Current or recent history (within the last six months) of alcohol or substance abuse.

Active infections or untreated systemic diseases that may interfere with the intervention or outcomes.

History of temporomandibular joint surgery or recent invasive dental procedures (within the last three months).

Known contraindications to TMS or tDCS, including intolerance to neuromodulation.

Participation in another clinical trial within the last three months.

Randomization

Participants will be randomly allocated to the control or intervention group by an independent investigator using an electronic randomization tool (Research Randomizer). Allocation will remain concealed until completion of assessments.

Sample Size Calculation

Sample size estimation indicates the need for 15 participants per group to ensure a statistical power of 85% (β = 0.20) and a significance level of p < 0.05. The final sample size was expanded to enhance the robustness of statistical analyses and to compensate for potential dropouts.

Assessment Instruments Visual Analogue Scale (VAS)

A 0-10 numerical scale used to quantify pain intensity, where 0 indicates no pain and 10 represents the worst imaginable pain.

Brief Pain Inventory (BPI)

A multidimensional tool that assesses pain intensity and pain interference with daily activities over the past 24 hours.

Graded Chronic Pain Scale (GCPS)

A scale that classifies chronic pain into severity grades based on pain intensity and functional disability.

SF-36 Health Survey

A generic quality-of-life questionnaire comprising 36 items distributed across eight domains, with scores ranging from 0 (worst health status) to 100 (best health status).

Manchester Orofacial Pain Disability Scale

An instrument that measures functional disability associated with orofacial pain, focusing on daily activities such as chewing and speaking.

Pressure Pain Threshold (PPT)

Assessed using a portable algometer. The minimum pressure that elicits a painful sensation will be recorded. Each site will be measured twice, and the mean value will be used for analysis.

Intervention Transcranial Direct Current Stimulation (tDCS)

tDCS will be administered using 35 cm² electrodes for 20 minutes across five consecutive days. The anode will be positioned at C3 or C4, contralateral to the primary site of pain, according to the international 10-20 EEG system. The control group will receive sham stimulation with identical electrode placement and procedures.

Transcranial Magnetic Stimulation (TMS)

TMS will be delivered in 10 sessions over two weeks. The intervention group will receive active stimulation, while the control group will receive sham stimulation. Stimulation parameters (frequency, intensity, and coil placement) will follow standardized clinical research guidelines for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants between 18 and 75 years old.
* Diagnosis of Chronic Orofacial Pain: Patients with persistent orofacial pain for more than 3 months, confirmed using DC/TMD or other validated diagnostic criteria.
* Pain Intensity: Baseline score on the Visual Analogue Scale (VAS) ≥ 4 (moderate to severe pain).
* Treatment History: Patients who have previously tried at least one conventional treatment (e.g., medication or physiotherapy) with limited or no success.
* Cognitive Ability: Participants cognitively able to understand the study procedures and provide informed consent.
* Stable Medication Regimen: Stable chronic pain medication for at least four weeks prior to the intervention.

Exclusion Criteria:

* Neurological Disorders: History of epilepsy, seizures, or other neurological disorders that contraindicate TMS or tDCS.
* Implanted Medical Devices: Presence of pacemakers, cochlear implants, or other electronic/metallic devices in the head or neck region.
* Pregnancy: Pregnant or breastfeeding individuals, due to potential risks.
* Psychiatric Disorders: Severe psychiatric disorders (e.g., schizophrenia, unstable major depression) that may interfere with study adherence.
* Substance Abuse: Current or recent history (within the last 6 months) of alcohol or substance abuse.
* Active Medical Conditions: Active infections or untreated systemic diseases that may interfere with results.
* TMJ Surgery: History of recent temporomandibular joint surgery or invasive dental procedures (within the last 3 months).
* Contraindications for TMS/tDCS: Sensitivity, intolerance, or inability to tolerate the neuromodulation device.
* Participation in Another Study: Simultaneous or recent (within the last 3 months) participation in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Assessed by Visual Analogue Scale (VAS) | Baseline, at the end of the 2-week intervention period (after 10 sessions), and 1 month after completion of the intervention
  Pain intensity will be assessed using a 10-cm Visual Analogue Scale (VAS), in which participants rate their average pain intensity by marking a point on a horizontal line anchored by "no pain" (0) and "worst pain imaginable" (10). Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Pain Interference Measured by the Brief Pain Inventory (BPI) | Baseline, at the end of the 2-week intervention period (after 10 sessions), and 1 month after completion of the intervention
  Pain-related interference will be evaluated using the interference subscale of the Brief Pain Inventory (BPI). The BPI assesses the extent to which pain interferes with daily activities, including general activity, mood, walking ability, work, relationships, sleep, and enjoyment of life. Each item is rated on a 0-10 numeric scale, with higher scores indicating greater interference.
Chronic Pain Severity Assessed by the Graded Chronic Pain Scale (GCPS) | Baseline, at the end of the 2-week intervention period (after 10 sessions), and 1 month after completion of the intervention
  Chronic pain severity will be assessed using the Graded Chronic Pain Scale (GCPS), which classifies pain according to pain intensity and pain-related disability. The GCPS generates grades ranging from Grade 0 (no pain) to Grade IV (high disability-severely limiting), with higher grades indicating greater pain-related impairment.
Health-Related Quality of Life Measured by SF-36 | Baseline, at the end of the 2-week intervention period (after 10 sessions), and 1 month after completion of the intervention
  Health-related quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36), which evaluates eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Scores for each domain range from 0 to 100, with higher scores indicating better perceived health status.
Pressure Pain Threshold (PPT) | Baseline, at the end of the 2-week intervention period (after 10 sessions), and 1 month after completion of the intervention
  Pressure pain threshold will be measured using a pressure algometer applied to predefined orofacial and/or cervical muscle sites. PPT is defined as the minimum pressure (expressed in kPa or kg/cm²) at which pressure sensation becomes painful. Higher PPT values indicate lower pain sensitivity.
Orofacial Functional Disability Assessed by the Manchester Orofacial Pain Disability Scale (MOPDS) | Baseline, at the end of the 2-week intervention period (after 10 sessions), and 1 month after completion of the intervention
  Orofacial functional disability will be evaluated using the Manchester Orofacial Pain Disability Scale (MOPDS), a self-reported questionnaire that assesses the impact of orofacial pain on daily functional activities. Higher scores reflect greater levels of functional disability related to orofacial pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health and Science, Almada, Setúbal District, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) from this study will not be shared with other researchers.
  Rationale for Non-Sharing:
  Informed Consent Limitations: The current informed consent forms signed by participants do not explicitly authorize the future public sharing or distribution of individual raw data, which limits our ability to comply with broad data sharing requests while maintaining ethical compliance.
  Data Sensitivity and Privacy: The collected data involves sensitive clinical information regarding chronic pain and psychiatric history. Although data is anonymized, the potential for re-identification, especially within small subgroups defined by specific conditions (e.g., both chronic orofacial pain and specific comorbidities), necessitates a conservative approach to protect participant privacy.
  Study Specificity: The complex, multi-modal intervention (TMS/tDCS) and assessment protocols used are highly specific to the research team's infrastructure and methodology, making the data

REFERENCES:
- [Background] Fricova J, Englerova K, Rokyta R. Noninvasive transcranial direct current stimulation (tDCS) for the treatment of orofacial pain. Neuro Endocrinol Lett. 2016 Oct;37(5):368-372. PMID 28231681
- [Result] Fricova J, Rokyta R. Transcranial Neurostimulation (rTMS, tDCS) in the Treatment of Chronic Orofacial Pain. Prog Neurol Surg. 2020;35:125-132. doi: 10.1159/000511134. Epub 2020 Oct 12. PMID 33045706
- [Result] Mayor RS, Ferreira NR, Lanzaro C, Castelo-Branco M, Valentim A, Donato H, Lapa T. Noninvasive transcranial brain stimulation in central post-stroke pain: A systematic review. Scand J Pain. 2024 Jul 3;24(1). doi: 10.1515/sjpain-2023-0130. eCollection 2024 Jan 1. PMID 38956966
- [Result] Olivieri G, Bodycote J, Wolff S. Adaptive response of human lymphocytes to low concentrations of radioactive thymidine. Science. 1984 Feb 10;223(4636):594-7. doi: 10.1126/science.6695170.
- [Result] Mizoguchi M, Omura Y, Hiyama T, Hirano H, Oka Y. [Combined resection of thyroid cancer with the common carotid artery and implantation of blood vessel prosthesis]. Iryo. 1967 May;21(5):585-91. No abstract available. Japanese. PMID 6078189
- [Result] Knotkova H, Hamani C, Sivanesan E, Le Beuffe MFE, Moon JY, Cohen SP, Huntoon MA. Neuromodulation for chronic pain. Lancet. 2021 May 29;397(10289):2111-2124. doi: 10.1016/S0140-6736(21)00794-7. PMID 34062145